CLINICAL TRIAL: NCT07244783
Title: Evaluation of the Effectiveness of a Web-Based Breastfeeding Education Program Based on the Information-Motivation-Behavioral Skills (IMB) Model
Brief Title: Effectiveness of an IMB Model-Based Web Breastfeeding Education Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ömür Aktaş, Sub-Investigator / Researcher, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-84892257-300-292373
Record Dates: First submitted 2025-08-18; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breastfeeding Education; Web Education
Keywords: Web-Based Breastfeeding Education; breast milk; breastfeeding; Information-Motivation-Behavioral Skills (IMB) Model
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in the IMB-based web breastfeeding education program (Active Comparator): This study evaluates a web-based breastfeeding education program structured according to the Information-Motivation-Behavioral Skills (IMB) model. The intervention group will receive a five-module program covering the importance of breastfeeding, breastfeeding techniques, common problems, mother-infant bonding, and stress management. The program includes educational texts, videos, digital guides, quizzes, and interactive tools. Motivation will be supported through virtual badges, motivational messages, and a certificate of participation. Behavioral skills will be assessed via web-based questionnaires and self-assessment scales.
  Interventions: Behavioral: Web-Based Breastfeeding Education Program
- Participants receiving routine hospital-based breastfeeding education (No Intervention): Participants in the control group will receive the standard hospital-based breastfeeding education routinely provided by healthcare professionals.

INTERVENTIONS:
Behavioral: Web-Based Breastfeeding Education Program — his study evaluates a web-based breastfeeding education program structured according to the Information-Motivation-Behavioral Skills (IMB) model. The intervention group will receive a five-module program covering the importance of breastfeeding.The program includes educational texts, videos, digital guides, quizzes, and interactive tools. Motivation will be supported through virtual badges, motivational messages, and a certificate of participation. Behavioral skills will be assessed via web-based questionnaires and self-assessment scales.
  Arms: Participants in the IMB-based web breastfeeding education program

SUMMARY:
This study is designed to evaluate the effectiveness of a Web-Based Breastfeeding Education Program based on the Information-Motivation-Behavioral Skills (IMB) Model. The study aims to examine the effects of the program on breastfeeding self-efficacy, motivation, problems encountered, and exclusive breastfeeding status among primiparous women.

Although breastfeeding is the most appropriate and natural form of infant nutrition, breastfeeding rates are still below the desired level both worldwide and in Turkey. According to the 2018 Turkey Demographic and Health Survey, breastfeeding is initiated at a high rate in the immediate postpartum period; however, continuation rates remain low. The main reasons for this include lack of maternal knowledge, limited social support, and restricted access to professional counseling. The recent increase in digital opportunities has introduced web-based interventions in breastfeeding education. Studies in the literature have shown that technology-assisted interventions improve maternal knowledge and motivation and contribute to sustaining breastfeeding.

In the first stage of this study, the Breastfeeding Knowledge Test (ASEBT) will be developed and its reliability assessed. The test, prepared based on a literature review and expert opinions, will consist of 30 multiple-choice questions. Reliability and validity analyses will be conducted using the KR-20 coefficient.

The second stage will be conducted as a randomized controlled trial. The sample will consist of 70 primiparous pregnant women who meet the inclusion criteria. Participants will be randomly assigned to intervention and control groups. The intervention group will receive a five-module web-based education program structured according to the IMB model. The modules will cover the importance of breastfeeding, breastfeeding techniques, common problems, mother-infant bonding, and stress management. The program will be supported with digital guides, mini quizzes, virtual badges, motivational messages, and achievement certificates. The control group will only receive routine hospital education.

Data will be collected using the Individual Information Form, ASEBT, Antenatal and Postnatal Breastfeeding Self-Efficacy Scales, Visual Analog Scale for Motivation, Breastfeeding Motivation Scale, Breastfeeding Problems Assessment Scale, and postpartum follow-up forms. All data will be analyzed using SPSS 22.0 software. After testing normality assumptions, descriptive statistics, independent sample t-tests, and Pearson correlation analyses will be applied. Results will be evaluated at a 95% confidence interval and a significance level of p<0.05.

Ethical approval and institutional permissions will be obtained prior to implementation. In addition, permissions for the use of the scales will be secured from the original authors. Participation will be voluntary, and informed consent will be obtained from all participants. Throughout the study, ethical principles including confidentiality, respect for autonomy, and non-maleficence/beneficence will be observed.

This study aims to introduce a digital-based approach to enhance behavioral outcomes related to breastfeeding. The web-based education program structured according to the IMB Model is expected to improve maternal knowledge and motivation, strengthen breastfeeding self-efficacy, and contribute to longer durations of exclusive breastfeeding. The study is anticipated to provide evidence to support the development and dissemination of technology-assisted educational programs in nursing practice.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of a Web-Based Breastfeeding Education Program based on the Information-Motivation-Behavioral Skills (IMB) Model among primiparous women. The research aims to assess the program's impact on breastfeeding self-efficacy, maternal motivation, breastfeeding-related problems, and exclusive breastfeeding rates.

Background

Although breastfeeding is universally recognized as the optimal and natural method of infant nutrition, both global and national rates remain below desired levels. According to the 2018 Turkey Demographic and Health Survey (TDHS), breastfeeding is initiated at high rates within the first hour postpartum; however, continuation of exclusive breastfeeding until six months remains limited. Key barriers include inadequate maternal knowledge, insufficient social support, and limited access to professional counseling. Nurses play a pivotal role in supporting breastfeeding through education and counseling, yet time constraints, limited staff availability, and accessibility challenges restrict face-to-face counseling. With the rapid expansion of digital technologies, web-based interventions have become promising alternatives for delivering breastfeeding education. Prior studies have shown that technology-assisted interventions improve maternal knowledge, motivation, and breastfeeding outcomes.

Objectives and Hypotheses

The primary objective of this study is to evaluate the effectiveness of a web-based breastfeeding education program structured according to the IMB Model. It is hypothesized that the program will improve maternal breastfeeding knowledge, motivation, self-efficacy, and exclusive breastfeeding rates while reducing breastfeeding-related problems compared to routine care.

Study Design

The study will be conducted in two phases:

Phase 1 - Development of the Breastfeeding Knowledge Test (ASEBT):

A 30-item multiple-choice test will be developed to assess breastfeeding knowledge.

Test items will be prepared based on literature review, Bloom's cognitive taxonomy, and expert consultation.

Content validity will be evaluated through expert review (n=9). The test will be administered to 300 pregnant women meeting the inclusion criteria.

Reliability will be assessed using the Kuder-Richardson (KR-20) coefficient; items with KR-20 below 0.60 will be excluded.

Phase 2 - Randomized Controlled Trial (RCT):

Sample and Randomization: A total of 80 primiparous pregnant women (≥32 weeks gestation, ≥19 years, literate, with access to internet-enabled devices) will be recruited from a university hospital's obstetrics outpatient clinic. Participants will be randomly assigned to intervention (n=35) and control (n=35) groups using a computer-generated randomization schedule. Exclusion criteria include mental or sensory impairments, psychiatric diagnoses, high-risk pregnancies, or prior structured breastfeeding education.

Intervention Group: Participants will complete a five-module web-based breastfeeding education program based on the IMB Model, which includes:

The Importance of Breastfeeding and Breast Milk

Understanding Infant Needs and Breastfeeding Techniques

Common Breastfeeding Problems and Management

Mother-Infant Bonding and Secure Attachment

Stress Management during the Breastfeeding Process The program incorporates interactive educational videos, digital breastfeeding guides, mini knowledge tests, motivational messages, virtual badges, and digital achievement certificates. Modules must be completed sequentially by 37 weeks of gestation.

Control Group: Participants will receive routine hospital-based breastfeeding education only. After study completion, the web-based program will be made available to the control group.

Follow-Up and Assessments:

Baseline (32-34 weeks): Individual Information Form, ASEBT (pre-test), Antenatal Breastfeeding Self-Efficacy Scale, Visual Analog Scale (VAS-Motivation).

37 weeks gestation: ASEBT (post-test), Antenatal Breastfeeding Self-Efficacy Scale, VAS-Motivation.

Within 48 hours postpartum: Postnatal Breastfeeding Self-Efficacy Scale, Breastfeeding Motivation Scale, Breastfeeding Problems Assessment Scale, Postpartum Follow-up Form 1.

1 month postpartum: ASEBT, Postnatal Breastfeeding Self-Efficacy Scale, Breastfeeding Motivation Scale, Breastfeeding Problems Assessment Scale, Postpartum Follow-up Form 2, exclusive breastfeeding status.

Data Collection Tools

Breastfeeding Knowledge Test (ASEBT) - developed in Phase 1. Antenatal and Postnatal Breastfeeding Self-Efficacy Scales Visual Analog Scale (VAS) for Motivation - to measure antenatal motivation. Breastfeeding Motivation Scale - adapted for Turkish mothers Breastfeeding Problems Assessment Scale - validated Turkish version Postpartum Follow-up Forms - developed based on current literature. Statistical Analysis

Data will be analyzed using SPSS 22.0. Normality will be tested prior to analysis. Descriptive statistics (mean, SD, frequency, percentage) will be calculated. Independent samples t-tests will be used to compare group means, and Pearson correlation will assess relationships between variables. Results will be evaluated at a 95% confidence interval with a significance level of p<0.05.

Ethical Considerations

Ethical approval have been obtained from Ankara Yıldırım Beyazıt University Ethics Committee and institutional permissions have been secured. Permissions for the use of all scales have been requested from the original authors. Participation will be voluntary, and written informed consent will be obtained from all participants. The principles of confidentiality, respect for autonomy, and beneficence/non-maleficence will be strictly observed.

Expected Contributions

This study is expected to provide evidence on the effectiveness of web-based, IMB model-guided breastfeeding education in improving maternal knowledge, motivation, and self-efficacy while reducing breastfeeding problems. By supporting exclusive breastfeeding practices, the intervention may contribute to improved maternal and child health outcomes. Findings are anticipated to guide the integration of technology-assisted interventions into routine nursing practice and to promote the wider dissemination of digital breastfeeding education programs.

ELIGIBILITY:
Inclusion Criteria (Second Phase of the Study)

Participants will be included if they meet all of the following criteria:

* Able to communicate in Turkish
* Literate (able to read and write)
* At 32 weeks of gestation or more
* Primiparous (first-time mother)
* Aged 19 years or older
* Have access to a device (smartphone or computer) with an internet connection, compatible with Android or iOS operating systems

Exclusion Criteria:

* Have conditions that may cause communication difficulties (e.g., mental, visual, or hearing impairments)
* Have a diagnosed psychiatric disorder (e.g., bipolar disorder, schizophrenia)
* Have a high-risk pregnancy (e.g., gestational diabetes, preeclampsia, multiple pregnancy, pregnancy after in vitro fertilization)
* Have previously received structured breastfeeding or breast milk education outside the hospital

Withdrawal Criteria:

Participants will be removed from the study if they meet any of the following:

* Choose to withdraw from the study at any stage
* Do not complete the web-based education modules after enrollment
* The newborn requires intensive care after birth
* The mother requires intensive care before or after birth

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding status: The proportion of infants exclusively receiving breast milk will be assessed in both the intervention and control groups at birth and at 1 month postpartum | The proportion of infants exclusively receiving breast milk will be assessed in both the intervention and control groups at birth and at 1 month postpartum
  The proportion of infants exclusively receiving breast milk will be assessed in both the intervention and control groups at birth and at 1 month postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.emzirmeyolculugu.com/

DOCUMENTS (1):
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT07244783/ICF_000.pdf